CLINICAL TRIAL: NCT06309732
Title: GAMEC-SHORT (S) & GAMEC-ANTHRACYCLINE(A) (Combination Chemotherapy With GCSF, Actinomycin-D, Methotrexate, Etoposide and Cisplatin) Risk-adapted Protocol for Relapsed Germ Cell Tumours (GCT)
Brief Title: GAMEC-II, Risk-adapted Protocol for Relapsed Germ Cell Tumours (GCT)
Acronym: GAMEC-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4491; 2006-001963-52 (EudraCT Number); TE 2006-09 (Other: Barts and the London NHS Trust)
Record Dates: First submitted 2014-09-09; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Testicular Neoplasms
Keywords: Germ cell tumour
MeSH Terms: conditions — Testicular Neoplasms; Neoplasms, Germ Cell and Embryonal | interventions — pegfilgrastim; Filgrastim; Dactinomycin; Methotrexate; Etoposide; etoposide phosphate; Cisplatin; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GAMEC - S (Experimental): Day 4 PEG Filgrastim 6mg Day 1 Actinomycin D 1mg/m2 Day 1 Methotrexate (dependent on creatinine clearance) Days 1,2, 3, 4 Etoposide 90mg/m2 Days 2, 3 Cisplatin 50mg/m2 Day 8 Cisplatin 50mg/m2 (cycle 1&2 only)
  Interventions: Drug: Dactinomycin; Drug: Methotrexate; Drug: Etoposide; Drug: Cisplatin
- GAMEC-A (Experimental): Day 1 Actinomycin-D 1m/m2 Day 2, 3 and 8 Methotrexate 8g/m2 (dependent on creatinine clearance) Day 2, 3 and 8 Cisplatin 50mg/m2 (Day 8 dose omitted from week 6 onwards) Day 1 and 2 Epirubicin 37.5mg/m2 Day 3 Pegfilgrastim 6mg Treatment given on weeks 1, 3, 6, 8 and 10.
  Interventions: Drug: Pegfilgrastim; Drug: Dactinomycin; Drug: Methotrexate; Drug: Cisplatin; Drug: Epirubicin

INTERVENTIONS:
Drug: Pegfilgrastim — 6mg at each cycle
  Other Names: Neupogen; Ratiograstim; Zarzio
  Arms: GAMEC-A
Drug: Dactinomycin — 1mg/m2
  Other Names: Cosmegen Lyovac
Drug: Methotrexate — Doses are titrated against renal function. Dosage: 30 mins loading plus 12 hour infusion
Drug: Etoposide — 90mg/m2 injection for infusion
  Other Names: Etopophos
  Arms: GAMEC - S
Drug: Cisplatin — 50mg/m2
Drug: Epirubicin — 37.5mg/m2
  Arms: GAMEC-A

SUMMARY:
St Bartholomew's hospital completed a study using the regimen GAMEC (PEG-filgrastim, actinomycin-D, methotrexate, etoposide, cisplatin). The results of this study showed that 50% of patients with relapsed testicular cancer could be cured using this treatment. These results are very encouraging and compare very favourably to other treatment protocols. In reviewing this study, it became clear that of the 5 cycles of treatment which were proposed, the first 3 seemed to matter and the last 2 did not appear important. In addition there was a group of patients who appeared to do particularly well namely patients under the age of 35 and those who had a normal LDH (lactate dehydrogenase). LDH is a blood test which monitors cancer activity. Selecting patients which fill both these criteria, this trial aims to see whether the investigators can maintain the good results the investigators have seen but using only 3 cycles of treatment. This will therefore shorten the treatment from 10 weeks to 6 weeks, thus reducing the side effects.

DETAILED DESCRIPTION:
GAMEC-II (GAMEC -S & GAMEC-A) is an open-labelled, non-randomised clinical trial in patients with relapsed germ cell tumours (GCT) and its objectives are:

1. To establish the response rates to GAMEC-S or GAMEC-A
2. To establish the safety and efficacy of substitution of epirubicin for etoposide (GAMEC-A regimen)
3. To establish the toxicity of GAMEC-A
4. To establish progression free survival (PFS)
5. To establish whether shortening GAMEC-S in patients without adverse prognostic factors reduces toxicity without compromising survival.

ELIGIBILITY:
Inclusion Criteria:

* Germ Cell Tumour (GCT), relapsed or progressing on or following platinum-based chemotherapy - as evidenced by rising tumour markers or progressive disease on CT scan
* Neutrophil count >1.0 x109/l
* Platelets >70 x109/l
* Haemoglobin >100g/l (may be transfused)
* Creatinine clearance should be >60ml/min. However, if creatinine clearance <60 ml/min then an EDTA clearance is MANDATORY. (If EDTA clearance is <60 ml/min then the patient will be excluded.)
* Males age >16 ≤35 years [decision made on physical fitness to participate]
* ECOG Performance status 0-3
* Full written consent

Exclusion Criteria:

* Other malignancy except basal cell carcinoma
* Evidence of clinically significant cardiac failure, unstable angina or uncontrolled hypertension
* Current participation in any other investigational drug study

Ages: 16 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Response rate to GAMEC-S or GAMEC-A | 6 weekly
  Tumour markers, clinical and radiological assessment of disease and/or examination of resected tissue (if surgery is done)

SECONDARY OUTCOMES:
Relapse-free survival | Monthly for 1 year, 2 monthly for 2nd year, 3 monthly 3rd year, annually there after
  CT-scan chest, abdomen and pelvis (continued pelvic scanning is dependent whether disease present)
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shamash, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts and the London NHS Trust, London, United Kingdom